CLINICAL TRIAL: NCT01495299
Title: 24-hour IOP Fluctuation Profile Recorded With SENSIMED Triggerfish in Primary Open-angle Glaucoma (POAG) Patients After Cataract Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Due to staff departures we were unable to execute this study
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: TDCAT1
Record Dates: First submitted 2011-12-12; First posted 2011-12-20 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Glaucoma
Keywords: relationship; IOP fluctuations; glaucoma; cataract surgery; SENSIMED Triggerfish
MeSH Terms: conditions — Glaucoma | interventions — Phacoemulsification; Lens Implantation, Intraocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cataract patients with glaucoma
  Interventions: Device: Phacoemulsification with implantation of intraocular lens (CE-IOL) SENSIMED Triggerfish

INTERVENTIONS:
Device: Phacoemulsification with implantation of intraocular lens (CE-IOL) SENSIMED Triggerfish — Phacoemulsification (standard cataract extraction surgery)

SUMMARY:
The purpose of this study is to determine the relationship between intraocular pressure (IOP) fluctuations of glaucoma patients as recorded with an IOP-sensing contact lens (SENSIMED Triggerfish®), during two 24-hour periods, before and after cataract surgery. This device has previously been investigated and shown to be safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to comply with the study procedures

  * 18-80 years old
  * Subjects diagnosed with glaucoma, based on presence of repeatable visual field loss and/or glaucomatous optic neuropathy based on masked review of optic disc stereophotographs and under ocular hypotensive treatment, or diagnosed with ocular hypertension, with an IOP of > 22 mmHg at the screening visit and under ocular hypotensive treatment.
  * Subject has consented to be in the trial
  * Visual acuity of 20/200 or better
  * Presence of cataract requiring phacoemulsification with lens exchange
  * Ability to understand the character and individual consequences of the study
  * For women of childbearing potential, adequate contraception

Exclusion Criteria:

* Subjects presenting with any of the following criteria will not be included in the trial:

  * Subjects with contraindications for wearing contact lenses
  * Severe dry eye syndrome
  * Keratoconus or other corneal abnormality
  * Conjunctival or intraocular inflammation
  * Eye surgery prior to and throughout the study.
  * Full frame metal glasses during SENSIMED Triggerfish® monitoring
  * Known hypersensitivity to silicone, plaster or ocular anesthesia (proparacaine)
  * Pregnancy and lactation
  * Simultaneous participation in other clinical studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: glaucoma patients scheduled to undergo cataract surgery.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
24-h IOP patterns | 24 hour

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD, La Jolla, California, United States